CLINICAL TRIAL: NCT01625897
Title: A Long-term Study of MP-214 in Patients With Chronic Phase or Elderly Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A002-A7
Record Dates: First submitted 2012-06-19; First posted 2012-06-22 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Mental Disorder; Psychotropic Drugs; Dopamine Agents; Risperidone; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Risperidone

ARMS (2):
- MP-214 1.5-9mg (Experimental)
  Interventions: Drug: MP-214
- Risperidone 2-12mg (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: MP-214 — Patients who meet eligibility criteria will be administered a once daily oral fixed dose (3mg or 6mg) of MP-214 for four weeks, then flexible dose (1.5-9mg) of MP-214
  Arms: MP-214 1.5-9mg
Drug: Risperidone — Patients who meet eligibility criteria will be administered a once daily oral fixed dose (4mg) of risperidone for two weeks, then flexible dose (2-12mg) of risperidone
  Arms: Risperidone 2-12mg

SUMMARY:
The objective of this study is to evaluate the long-term safety, tolerability, and efficacy of MP-214 in patients with chronic phase or elderly schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient before the initiation of any study-specific procedures
* Patients diagnosed with schizophrenia according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia
* Patients who meet at least one of the following:

  * current diagnosis of schizophrenia of chronic phase
  * between 65 and 74 years of age
* Patients with normal physical examination, laboratory, vital signs, and/or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of schizoaffective disorder, schizophreniform disorder, other psychotic disorders other than schizophrenia, or bipolar I or II disorder

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aizu-Wakamatsu, Fukushima, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-214 1.5-9mg: Patients who meet eligibility criteria will be administered a once daily oral fixed dose (3mg or 6mg) of MP-214 for four weeks, then flexible dose (1.5-9mg) of MP-214
- Risperidone 2-12mg: Patients who meet eligibility criteria will be administered a once daily oral fixed dose (4mg) of risperidone for two weeks, then flexible dose (2-12mg) of risperidone
Period: Overall Study
Arm/Group | MP-214 1.5-9mg | Risperidone 2-12mg
Started | 83 | 42
Completed | 31 | 28
Not Completed | 52 | 14
Not completed — Adverse Event | 27 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 25 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-214 1.5-9mg | Risperidone 2-12mg | Total
Number analyzed (Participants) | 83 | 42 | 125
Age, Customized [Count of Participants; unit: Participants]
  >=20 and <65 years | 66 | 32 | 98
  >=65 and <74 years | 17 | 10 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 18 | 62
  Male | 39 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: Up to 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MP-214 1.5-9mg | Risperidone 2-12mg
Number analyzed (Participants) | 83 | 42
Participants | 78 | 42

ADVERSE EVENTS:
Arm/Group | MP-214 1.5-9mg | Risperidone 2-12mg
Serious Adverse Events (participants affected / at risk) | 13/83 | 4/42
Other Adverse Events (participants affected / at risk) | 72/83 | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 1.5-9mg (N=83) | Risperidone 2-12mg (N=42)
Cholangitis (Hepatobiliary disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 9 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 1.5-9mg (N=83) | Risperidone 2-12mg (N=42)
Hyperprolactinaemia (Endocrine disorders) | 6 | 16
Constipation (Gastrointestinal disorders) | 7 | 3
Dental caries (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 15 | 5
Vomiting (Gastrointestinal disorders) | 8 | 3
Malaise (General disorders) | 3 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 0
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 26 | 14
Blood creatine phosphokinase increased (Investigations) | 8 | 4
Blood prolactin increased (Investigations) | 9 | 12
Blood urine present (Investigations) | 5 | 1
Weight increased (Investigations) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Akathisia (Nervous system disorders) | 5 | 8
Headache (Nervous system disorders) | 5 | 5
Parkinsonism (Nervous system disorders) | 2 | 6
Somnolence (Nervous system disorders) | 8 | 5
Insomnia (Nervous system disorders) | 14 | 12
Schizophrenia (Nervous system disorders) | 28 | 11
Suicidal ideation (Nervous system disorders) | 3 | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3
Hypertension (Vascular disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other